CLINICAL TRIAL: NCT03945214
Title: Program on Work Stress and Health Outcomes in a Heterogeneous University Employee Cohort
Brief Title: The Impact of 8 Weeks of Digital Meditation Application and Healthy Eating Program on Work Stress and Health Outcomes
Acronym: SFUC+Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The University of California's Healthy Campus Network (Other); Headspace, Inc (Unknown); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 17-23717-2; K23AT011048-01 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Stress; Psychological; Behavioral Symptoms; Sleep; Health Behavior; Weight, Body
Keywords: Stress; Health; Meditation; Eating; Mindfulness; Employees; Job strain; Burnout; Work; Mood; Affect; Work related stress; Blood pressure; Inflammation
MeSH Terms: conditions — Behavioral Symptoms; Health Behavior; Body Weight; Occupational Stress; Burnout, Psychological; Inflammation | interventions — Meditation; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Randomization to one of 4 conditions:
  1. Digital meditation condition
  2. Healthy eating condition
  3. Digital meditation + healthy eating condition
  4. Wait-list control
Who Masked: Investigator
Masking Description: Investigator will be blind to condition throughout data accrual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meditation group (Experimental): Participants in the meditation intervention group will be assigned to a digitally-based meditation intervention (Headspace app- Basics + Stress packs) and asked to use this for at least 10 minutes a day over the course of 8 weeks.
  Interventions: Behavioral: Meditation
- Healthy eating group (Experimental): Participants in the healthy eating group will be required to attend an in-person 50-minute counseling session geared towards developing goals to improve eating behavior, along with three 10-minute booster phone calls at weeks 1, 4, and 8. They will be asked to engage with a digital-based mindful eating program once per week over the course of 8 weeks.
  Interventions: Behavioral: Healthy Eating
- Mediation + Healthy eating group (Experimental): Participants in the meditation + healthy eating intervention group will be assigned to a digitally-based meditation intervention (Headspace app- Basics + Stress packs) and asked to use this for at least 10 minutes a day over the course of 8 weeks. They will also be required to attend an in-person 50-minute counseling session geared towards developing goals to improve eating behavior, along with three 10-minute booster phone calls at weeks 1, 4, and 8. They will be asked to engage with a digital-based mindful eating program once per week over the course of 8 weeks.
  Interventions: Behavioral: Meditation + healthy eating
- Waitlist control condition (No Intervention): Waitlist control group participants will continue their normal activities and not add any form of mediation during the study period.

INTERVENTIONS:
Behavioral: Meditation — 10 minute per day, 8 week digital meditation
  Arms: Meditation group
Behavioral: Healthy Eating — A single 50 minute counseling session focused on eating behaviors, and three 10-minute follow-up phone calls to check-in on eating goals
  Arms: Healthy eating group
Behavioral: Meditation + healthy eating — 10 minute per day, 8 week digital meditation and a single 50 minute counseling session focused on eating behaviors, and three 10-minute follow-up phone calls to check-in on eating goals
  Arms: Mediation + Healthy eating group

SUMMARY:
The aim of the present study is to test the effects of a digital meditation intervention and/or a healthy eating intervention in a sample of UCSF employees with overweight and obesity (BMI>=25kg/m2) who report mild to moderate stress. We will randomize UCSF employees to 8-weeks of a digital meditation intervention (using the commercially available application, Headspace), a healthy eating intervention, a digital meditation+healthy eating intervention, or a waitlist control condition.

DETAILED DESCRIPTION:
The aim of the present study is to test the effects of a digital meditation intervention and/or a healthy eating intervention in a sample of UCSF employees with overweight and obesity (BMI>=25kg/m2) who report mild to moderate stress. We will randomize UCSF employees to 8-weeks of a digital meditation intervention (using the commercially available application, Headspace), a healthy eating intervention, a digital meditation+healthy eating intervention, or a waitlist control condition.

Participants assigned to the digital meditation intervention group will be asked to download and use the Headspace mobile application for at least 10 minutes per day for 8 weeks. Participants assigned to the healthy eating intervention group will be asked to participate in a 50 minute motivational interviewing counseling session centered around healthy eating behaviors , three 10-minute booster phone calls at weeks 1, 4, and 8, and weekly participation in a digital mindful eating activity.

All study participants will be asked to fill out questionnaires at baseline, week 4, week 8 (post-intervention), and a 4-month follow-up period. Among participants who are randomized to the digital meditation intervention, they will also take part in a 1-year follow-up assessment. Physiological assessments (body composition, blood spot) will be obtained at an in-person clinic visit at baseline and week 8. Fitness, sleep, and mood data will be gathered for seven consecutive days at baseline and week 8.

Prior to randomization, participants will go through an eligibility screening and complete the baseline questionnaire battery. Adherence in the digital meditation intervention will be tracked remotely. The goal is to recruit up to 165 participants

ELIGIBILITY:
Inclusion Criteria:

You may join if you

* Have access to a smartphone or computer every day
* Are fluent in English
* Are a UCSF employee
* Report mild to moderate levels of stress (as determined by a Perceived Stress Scale score of 15 or higher)
* Consent: demonstrate understanding of the study and willingness to participate as evidenced by voluntary informed consent and have received a signed and dated copy of the informed consent form
* Are at least 18 years of age
* Express a willingness to be randomly assigned into the waitlist group or the intervention groups
* Report a Body Mass Index (BMI) of 25 kg/m2 or above

Exclusion Criteria:

You may not join if you:

* Are an experienced meditator or have participated in a formal meditation practice in the last 3 months (defined as 3 times per week or more for 10 minutes or more at each practice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-05-19 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aric Prather, PhD, Principal Investigator — UC San Francisco; Elissa Epel, PhD, Principal Investigator — UC San Francisco; Rachel Radin, PhD, Principal Investigator — UC San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radin RM, Epel ES, Mason AE, Vaccaro J, Fromer E, Guan J, Prather AA. Impact of digital meditation on work stress and health outcomes among adults with overweight: A randomized controlled trial. PLoS One. 2023 Mar 1;18(3):e0280808. doi: 10.1371/journal.pone.0280808. eCollection 2023. PMID 36857330

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Started | 39 | 41 | 41 | 42
Completed | 36 | 37 | 34 | 38
Not Completed | 3 | 4 | 7 | 4
Not completed — Lost to Follow-up | 3 | 4 | 7 | 4

BASELINE CHARACTERISTICS:
Population: Please note that while 163 participants were originally randomized, our total sample for analysis at baseline was 161 participants. This discrepancy is due to the discovery that 2 of the randomized participants were actually ineligible for the study (BMI was <25 kg/m2 when measured in person).
Groups:
- Total: Total of all reporting groups
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition | Total
Number analyzed (Participants) | 38 | 41 | 40 | 42 | 161
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 39 | 40 | 42 | 158
  >=65 years | 1 | 2 | 0 | 0 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.63 (11.01) | 39.29 (12.43) | 35.40 (8.03) | 38.33 (12.55) | 37.92 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 34 | 27 | 28 | 116
  Male | 11 | 7 | 13 | 14 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 6 | 2 | 20
  Not Hispanic or Latino | 31 | 36 | 34 | 40 | 141
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 7 | 8 | 13 | 32
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 3 | 4 | 5 | 3 | 15
  White | 23 | 19 | 20 | 22 | 84
  More than one race | 4 | 7 | 7 | 4 | 22
  Unknown or Not Reported | 2 | 4 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 40 | 42 | 161

OUTCOME MEASURES:

1. Primary Outcome: Change in Perceived Stress Score, as Determined by the Total Score on the Perceived Stress Scale
Description: The Perceived Stress Scale has a total score scale range of 0 to 40, with higher values indicating more perceived stress
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 144 total participants completed both baseline and follow-up (8 week) measures of PSS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 36 | 37 | 33 | 38
units on a scale | -5.972 (0.944) | -2 (0.931) | -4.97 (0.986) | -1.658 (0.919)

2. Primary Outcome: Change in Food Action and Acceptance and Action Questionnaire (FAAQ), as Determined by the Summary Score on the FAAQ
Description: The Food Acceptance and Action Questionnaire has a total score scale range of 10 to 60, with higher scores indicating greater acceptance of motivations to eat.
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 136 total participants completed both baseline and follow-up (8 week) measures of the FAAQ.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 35 | 35 | 29 | 37
units on a scale | 0.257 (1.372) | 1.8 (1.372) | -0.828 (1.507) | 0.8108 (1.334)

3. Secondary Outcome: Change in Work Overcommitment, as Determined by Siegrist Job Strain Scale (Effort-Reward Imbalance Scale)
Description: The job strain- overcommitment measure (6 items) has items ranging from 1 to 4 (total score ranges from 6-24). The job strain-overcommitment score is calculated as the sum of items 17-22, with higher scores reflecting greater likelihood of experiencing over-commitment at work..
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 139 total participants completed both baseline and follow-up (8 week) measures of Work Overcommitment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 33 | 36 | 33 | 37
units on a scale | -1.576 (0.534) | -1.056 (0.512) | -2.242 (0.534) | -0.054 (0.505)

4. Secondary Outcome: Change in Subjective Mindfulness, as Determined by Total Score on the Mindful Attention Awareness Scale
Description: The Mindful Attention Awareness Scale is a 15-item measure with each item ranging from a score of 1 to 6. To score the scale, we compute the average score across items, with a higher score reflecting higher levels of mindfulness.
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 132 total participants completed both baseline and follow-up (8 week) measures of the MAAS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 32 | 34 | 29 | 37
units on a scale | 0.508 (0.116) | 0.253 (0.112) | 0.423 (0.122) | -0.013 (0.108)

5. Secondary Outcome: Change in the Intentional Use of Palatable Food to Cope With Negative Feelings, as Determined by Total Score on the Palatable Eating Motives, Coping Subscale (PEMS)
Description: The Palatable Eating Motives, Coping Subscale is a 4-item measure, with each item ranging from 1 (almost never/never) to 5 (almost always/always). A total coping sub scale score is determined by an average of the 4 items. Higher scores reflect greater use of palatable food to cope with negative emotions.
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 133 total participants completed both baseline and follow-up (8 week) measures of the PEMS.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 31 | 34 | 31 | 37
units on a scale | -0.573 (0.168) | -0.044 (.16) | -0.339 (.168) | -0.135 (.154)

6. Secondary Outcome: Change in Food Cravings, as Determined by Total Score on the Trait Food Craving Questionnaire, Reduced (FCQ-T-r)
Description: The Trait Food Craving Questionnaire, reduced, is a 15-item measure of behavioral, cognitive, and physical aspects of cravings for different types of food. Item response choices range from 0 (never) to 5 (always), and the total score is a sum of the 15 items (total score ranges from 0-75). Higher scores reflect greater cravings to eat densely caloric snack.
Time Frame: Baseline to post-intervention, an anticipated average of 8 weeks
Population: Please note that while 163 participants were originally randomized, 2 of those individuals were found to be ineligible post-randomization (due to BMI being measured <25 kg/m2 during in-person visit). Furthermore, of the 161 participants included in baseline analyses, only 129 total participants completed both baseline and follow-up (8 week) measures of the FCQ-T-r.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
Number analyzed (Participants) | 30 | 33 | 29 | 37
units on a scale | -9 (1.926) | -5.939 (1.836) | -7.483 (1.959) | -4.378 (1.734)

ADVERSE EVENTS:
Time Frame: 1 year
Description: They do not differ.
Arm/Group | Meditation Group | Healthy Eating Group | Mediation + Healthy Eating Group | Waitlist Control Condition
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/41 | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/41 | 0/42
Other Adverse Events (participants affected / at risk) | 0/39 | 0/41 | 0/41 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT03945214/Prot_SAP_000.pdf